CLINICAL TRIAL: NCT06820996
Title: Effect of Cryotreated Sodium Hypochlorite Irrigation At Different Consentrations in Mandibular First Molars with Symptomatic Irreversible Pulpitis: a Randomized Controlled Trial
Brief Title: Effect of Cryotreated Sodium Hypochlorite Irrigation At Different Consentrations in Mandibular First Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Kübra Gürler, Cukurova University, Faculty of Dentistry, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 13.02.2025/150
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Pulpitis - Irreversible
Keywords: Cryotherapy; Irreversible pulpits; Sodium hypochlorite; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cryotreated %2.5 NaOCl (Experimental): A total of 45 ml of 2.5% NaOCl cooled to 2 °C in the refrigerator was placed in 2.5 ml syringes. The syringes were placed in a cold storage box to maintain the temperature during use. The box was filled with ice and the temperature was verified at 2 °C with a digital thermometer. During the root canal preparation, each canal was irrigated with a total of 10 ml of 2.5% NaOCl at 2 °C. The procedure was completed by using 5 ml of 2.5% NaOCl at 2.5 °C, 2 ml of saline, 2 mL of 17% EDTA and 2 ml of saline for each root canal, respectively, as the final irrigation solution.
  Interventions: Other: Cryotherapy
- Normal %2.5 NaOCl (Experimental): 45 milliliters (ml) of 2.5% NaOCl was placed in a glass container at room temperature and the temperature was monitored with a digital thermometer to ensure that it remained at 25 °C. During root canal preparation, each canal was irrigated with a total of 10 ml of 25 °C 2.5% NaOCl. The procedure was completed by using 5 ml of 25 °C 2.5% NaOCl, 2 ml of saline, 2 ml of 17% EDTA and 2 ml of saline for each root canal, respectively, as the final irrigation solution.
  Interventions: Other: Control (Standard treatment)
- Cryotreated %5 NaOCl (Experimental): A total of 45 ml of 5% NaOCl cooled to 2 °C in the refrigerator was placed in 2.5 ml syringes. The syringes were placed in a cold storage box to maintain the temperature during use. The box was filled with ice and the temperature was verified at 2 °C with a digital thermometer. During the root canal preparation, each canal was irrigated with a total of 10 ml of 5% NaOCl at 2 °C. As the final irrigation solution, 5 ml of 5% NaOCl at 2 °C, 2 ml of saline, 2 mL of 17% EDTA and 2 ml of saline were used for each root canal, respectively, to complete the procedure.
  Interventions: Other: Cryotherapy
- Normal %5 NaOCl (Experimental): 45 ml of 5% NaOCl was placed in a glass container at room temperature and the temperature was monitored with a digital thermometer to ensure that it remained at 25 °C. During the root canal preparation, each canal was irrigated with a total of 10 ml of 25 °C 5% NaOCl. As the final irrigation solution, 5 ml of 25 °C 5% NaOCl, 2 ml of saline, 2 ml of 17% EDTA and 2 ml of saline were used for each root canal, respectively, and the procedure was completed.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: Cryotherapy — The root canals were irrigated with 2 °C NaOCl solution in cryotherapy group.
  Other Names: Normal
  Arms: Cryotreated %2.5 NaOCl; Cryotreated %5 NaOCl
Other: Control (Standard treatment) — The root canals were irrigated with 25 °C NaOCl solution in normal group.
  Arms: Normal %2.5 NaOCl; Normal %5 NaOCl

SUMMARY:
The goal of this clinical trial was to evaluate the effect of cryotreated sodium hypochlorite solution on the intensity of postoperative pain in root canal treatment procedures in mandibular first molar teeth with symptomatic irreversible pulpitis. The main question it aims to answer is:

- Does controlled irrigation with cold sodium hypochlorite in root canal treatment reduce the severity of postoperative pain? In the cryotreated NaOCl group, unlike the normal NaOCl group, the root canals were irrigated with 2 °C NaOCl solution.

DETAILED DESCRIPTION:
Various irrigation solutions that are effective for organic and inorganic tissues are used during root canal treatment. Sodium hypochlorite (NaOCl) is the most commonly used irrigation solution. It has antibacterial and physicochemical properties 20 and is unique in dissolving organic tissues 21. NaOCl irrigation combined with mechanical instrumentation has been consistently shown to substantially reduce the microorganism load in root canals 22. There have been several attempts to increase the antimicrobial efficacy of NaOCl in the root canal system, such as changing its concentration, increasing the contact time with the dentin walls of the root canal, increasing the total volume of irrigation, increasing its temperature, and using manual or mechanical activation methods 3, 23. These methods to increase the efficacy of NaOCl can also result in heightened toxic effects on periapical tissues owing to the tissue-irritating properties of the solution. This extrusion into the periapical region increases postoperative pain, especially in teeth with open apices and necrotic pulps 21, 24. Therefore, instead of using high concentrations of NaOCl, which could increase its toxic effects, safer means, such as increasing its temperature and using it in large volumes, may increase its efficacy 21, 25.

Therefore, ascertaining the clinical impact of cryotreated NaOCl on postoperative pain is essential. The temperature of the irrigation solution is known to affect postoperative pain, and final irrigation with cold saline significantly reduces postoperative pain levels 19, 26. However, studies investigating the effects of cryotreated NaOCl, which is used in all stages of root canal treatment, and using NaOCl at concentrations of 2.5% and 5% on postoperative pain are lacking. This randomized clinical trial investigated the effects of cryotreated 2.5% and 5% NaOCl on postoperative pain during endodontic treatment procedures in mandibular first molars with symptomatic irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:• Vital mandibular first molars with 3 root canals that responded positively to the cold test and electric pulp test

* Mandibular first molars with a preoperative VAS value of 4 and above (no pain (0 mm), mild pain (1-3 mm), moderate pain (4-6 mm), severe pain (7-10 mm))
* Teeth without periapical radiolucency seen radiographically
* Patients who did not take analgesics or antibiotics in the last 24 hours before the procedure were included in the study.

Exclusion Criteria:

* Devital teeth that responded negatively to cold tests and electric pulp tests,
* Teeth with poor periodontal status (pocket depth > 4 mm),
* Mandibular first molars with 4 or more root canals detected radiographically or after opening the endodontic access cavity,
* Teeth with no preoperative pain or with mild preoperative pain (VAS value below 4) were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | up to 72 hours
  The visual analog scale for pain is a straight line with one end meaning no pain (0) and the other end meaning the worst pain (10) imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine. Also called VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Koray Yılmaz, DDS MSc, Principal Investigator — Cukurova Univercity
Locations (1):
- Cukurova University, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nandakumar M, Nasim I. Effect of intracanal cryotreated sodium hypochlorite on postoperative pain after root canal treatment - A randomized controlled clinical trial. J Conserv Dent. 2020 Mar-Apr;23(2):131-136. doi: 10.4103/JCD.JCD_65_20. Epub 2020 Nov 5. PMID 33384483
- [Background] Lalfakawmi S, Gupta A, Duraisamy AK, Abraham D, Mrinalini M, Mane AP. Impact of Cryotreated and Warm Sodium Hypochlorite on Postoperative Pain in Teeth With Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial. J Endod. 2024 Nov;50(11):1543-1550. doi: 10.1016/j.joen.2024.07.002. Epub 2024 Jul 8. PMID 38987018